CLINICAL TRIAL: NCT01911910
Title: Heart Attack Prevention Programme for You (HAPPY) London
Acronym: HAPPYLondon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Steffen Erhard Petersen, Reader in Advanced Cardiovascular Imaging, Honorary Consultant Cardiologist, Centre Lead for Advanced Cardiovascular Imaging, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ReDa: 007711
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Disease
Keywords: primary prevention; Cardiovascular disease; Cardiovascular magnetic resonance (CMR); Electronic coaching (e-coaching)
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Usual care that would be provided by the NHS Health Check or equivalent.
- Electronic coaching plus standard care (Experimental): Tailored coaching for participants randomised to use the HAPPY e-coaching tool. Access to lifestyle and heart health scores and personalised advice to improve suboptimal behaviour.
  Interventions: Behavioral: Electronic coaching plus standard care

INTERVENTIONS:
Behavioral: Electronic coaching plus standard care — The HAPPY London web-based tool will provide the participant with an individualised score for their lifestyle and 10 year CV risk score, based mainly on the modified Framingham score, and provide tailored advice and education on the suboptimal factors. Ideal targets will be set and the information will be updated at 3 and 6 months allowing the participant to view their progress. Weekly emails with brief health and lifestyle advice will be sent to encourage healthier behaviour based on clinical studies or topical issues in the media. Links to social networks, such as Facebook posting and the ability to allow chosen family and friends to view their progress will aim to further encourage healthier behaviour.
  Other Names: Electronic coaching; E-Coaching; HAPPY E-Coaching
  Arms: Electronic coaching plus standard care

SUMMARY:
Diseases of the heart and blood vessels, such as heart attacks and strokes, are very common and can lead to severe disability or death. Changes in the body leading to heart attacks and strokes usually develop over decades as a result of smoking, diet, and lack of exercise, obesity, diabetes and high blood pressure. Changes in lifestyle and diet can significantly reduce the risk of heart diseases. General Practitioners invite 40 to 74 year-olds who have no known heart disease to take part in the NHS Health Check, which measures each person's individual risk of developing a heart attack or stroke and encourages them in a face-to-face meeting to take part in programmes to help them to give up smoking, lose weight etc. where necessary. In this new clinical trial the investigators will test whether computer-tailored electronic (e)-coaching via email and the internet can help people make the necessary changes in their lifestyle to reduce the risk of heart attacks and strokes.

DETAILED DESCRIPTION:
Heart Attack Prevention Programme for You London (HAPPY London) will be conducted as a randomised controlled trial comparing the use of tailored e-coaching in addition to the standard of care vs. standard care alone. Standard care is defined as the care that would be offered by the NHS Health Check programme through the NHS primary care. We will use a range of established and novel cardiovascular markers to determine the clinical and cost effectiveness of e-coaching and gain pathophysiological insight into how lifestyle modifications affect the cardiovascular system. These measures include cardiovascular magnetic resonance imaging (CMR), aortic stiffness parameters, vascular ultrasound and other biomarkers of CV disease risk.

Intervention

The HAPPY London web-based tool will provide the participant with an individualised score for their lifestyle and 10 year CV risk score, based on the modified Framingham score and the UK specific QRisk Score, and provide tailored advice and education on the suboptimal factors. Ideal targets will be set and the information will be updated at 3 and 6 months allowing the participant to view their progress. Weekly emails with brief health and lifestyle advice will be sent to encourage healthier behaviour based on clinical studies or topical issues in the media. Links to social networks, such as Facebook posting and the ability to allow chosen 'buddies' from family or friends to view their progress will aim to further encourage healthier behaviour.

The study involves the recruitment of 400 adults between the age of 40 and 74 years who have a moderate to high 10-year CV risk score (Estimated 10 year CV risk >10%). Half of the study group will receive use of the e-coaching in addition to standard care allocated randomly stratified according to either moderate (QRisk between 10 and 20%) or high risk (QRisk more than or equal to 20%). The initial screening will take place on the www.happylondon.info web-based 'mini-check' questionnaire. Potential participants will then be seen at a physical screening visit to confirm eligibility. 3 subsequent visits will take place over 6 months; baseline, 3 month and 6 month follow up. A subgroup of the study population (65 from each intervention arm thus totalling 130 participants ) will also have a baseline and follow up cardiovascular magnetic resonance (CMR) imaging. Assessment will be performed using a variety of measures through questionnaires, blood pressure (BP) checks, blood tests, ultrasound scans, oscillometric method to assess pulse wave velocity and pulse wave analysis and CMR multi-parametric scanning.

The primary aim of this study is to assess the clinical effectiveness of individualised, continuous electronic (e-) coaching to support a healthier lifestyle as a primary prevention tool to reduce the CV risk and improve the quality of life in asymptomatic individuals with intermediate to high 10 year CV risk.

Other questions that we aim to answer are:

1. Is computer-tailored e-coaching cost-effective in the short-term (clinical trial period) and during the long-term (decision analysis modelling)
2. What are the associations of personality traits, economic preferences, and sociocultural factors with the achieved lifestyle modifications and changes in the cardiovascular phenotype?
3. What is the relationship between changes observed in markers derived from our multi-parametric cardiovascular magnetic resonance imaging protocols following lifestyle changes?
4. How frequent are silent myocardial infarctions in a typical NHS Health Check population?
5. Do treatment effects differ between ethnic groups?

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be enrolled following an informed consent. The subject will be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* Subjects will be between 40 and 74 years of age
* Subjects will have unrestricted access to the Internet
* Subjects will be sufficiently fluent in English language.
* Subjects will have an estimated intermediate to high risk for CV events based on the web-based pre-screening tool (www.happylondon.info), which is based on the nonlaboratory Framingham risk score (>10% 10 year cardiovascular risk)

Exclusion Criteria:

* History of stroke or transient ischaemic attack (TIA)
* Cardiac sounding chest pain requiring further investigations
* Current life threatening conditions other than vascular disease (e.g. very severe chronic airways disease, HIV positive, life-threatening arrhythmias) that may prevent a subject from completing the study
* Only for subgroup undergoing cardiac contrast-enhanced magnetic resonance studies: Any contraindication to a contrast-enhanced magnetic resonance study, such as known allergies to gadolinium-based contrast agents, severe claustrophobia, pacemakers, defibrillators, etc

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen E Petersen, MD DPhil, Principal Investigator — Queen Mary University of London
Locations (1):
- Centre for Advanced Cardiovascular Imaging, William Harvey Research Institute, Queen May University of London, London, United Kingdom

REFERENCES:
- [Result] Khanji MY, Balawon A, Boubertakh R, Hofstra L, Narula J, Hunink M, Pugliese F, Petersen SE. Personalized E-Coaching in Cardiovascular Risk Reduction: A Randomized Controlled Trial. Ann Glob Health. 2019 Jul 12;85(1):107. doi: 10.5334/aogh.2496. PMID 31298823
- [Derived] Khanji MY, Stone IS, Boubertakh R, Cooper JA, Barnes NC, Petersen SE. Chronic Obstructive Pulmonary Disease as a Predictor of Cardiovascular Risk: A Case-Control Study. COPD. 2020 Feb;17(1):81-89. doi: 10.1080/15412555.2019.1694501. Epub 2019 Dec 13. PMID 31833441

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Started | 197 | 205
Completed | 184 | 194
Not Completed | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care | Total
Number analyzed (Participants) | 197 | 205 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (4.8) | 65.1 (6.3) | 65.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 78 | 149
  Male | 126 | 127 | 253

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulse Wave Velocity (PWV)
Description: Change in aortic stiffness using a Vicorder device measured in m/s
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
m/s | -0.25 (1.73) | -0.16 (1.25)

2. Secondary Outcome: Change in Carotid Intima Media Thickness CIMT
Description: carotid intima media thickness CIMT as measured by ultrasound
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
mm | 0.01 (0.09) | 0.01 (0.08)

3. Secondary Outcome: Change in Quality of Life
Description: Lifestyle, quality of life and physical activity questionnaires. Questionnaires SF-36, EQ5D-3L, RPAQ.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Data not reported as full analysis not done due to time constraints
Population: Change in quality of life using the visual analogue scale (VAS) from the EQ-5D questionnaire. Not all participants completed both the baseline and 6-month follow-up, therefore resulting in a lower number analysed compared to other quantitative measures.The highest VAS is score was 1 (best values, highest quality of life).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 162 | 166
score on a scale | 0.01 (0.06) | 0 (0.16)

4. Secondary Outcome: Pulse Wave Velocity by CMR
Description: Change in aortic stiffness as measured by CMR derived aortic pulse wave velocity measured in m/s
Time Frame: Baseline and 6 month. Data not reported as full analysis not possible due to time and resource limitations.
Reporting Status: Not Posted, anticipated posting 2023-12

5. Secondary Outcome: Aortic Distensibility by Cardiovascular Magnetic Resonance (CMR)
Description: CMR will be performed on 65 participants in the treatment and 65 in the standard care group.
  Change in aortic stiffness - aortic distensibility (mmHg-1, CMR)).
Time Frame: Baseline and 6 month
Reporting Status: Not Posted

6. Secondary Outcome: Left Ventricular Mass by CMR
Description: Change in LV mass index (g/m2, CMR).
Time Frame: Baseline and 6 month
Population: CMR data were collected as part of a pilot data in a subgroup of the total number of participants enrolled in the study. Further analysis will take place once funding for further fellow who will be able to perform the detailed software analysis. The data will forms ongoing work.
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 42 | 44
g/m2 | -1.42 (8.36) | -1.73 (9.4)

7. Secondary Outcome: Left Ventricular Ejection Fraction by CMR
Description: LV end-diastolic and end-systolic volume indices, (ml/m2, CMR), LV EF (%, CMR).
Time Frame: Baseline and 6 month
Population: Change in the ejection fraction based on the moving images derived from the CMR scan.
Measure: Mean (Standard Deviation); unit: % change in ejection fraction
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 42 | 44
% change in ejection fraction | -0.45 (5.41) | -0.88 (6.29)

8. Secondary Outcome: Myocardial Fibrosis by CMR
Description: Extent and change in diffuse myocardial fibrosis (extracellular volume fraction measured as a %, derived from CMR imaging)
Time Frame: Baseline and 6 month. Baseline and 6 month. Data not reported as full analysis not possible due to time and resource limitations.
Reporting Status: Not Posted, anticipated posting 2023-12

9. Secondary Outcome: Diastolic Function by CMR
Description: Diastolic function (strain and strain rate in % and s-1, respectively derived from CMR imaging data).
  This is a measure of how stiff the main chamber of the heart is. The software to analyse these data will be available in the future.
  The raw images from the scan will be used for future analysis once software for this assessment is developed. Our group is working on developing this tool.
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2023-12

10. Secondary Outcome: Change in Framingham Risk Score
Description: Assessment of cardiovascular risk based on the Framingham algorithm. Minimum value 0% and maximum value theoretically 100%. Higher score means worse predicted outcome.
  Assessment of 10-year cardiovascular risk score based on the Framingham population derived algorithm.
  Minimum value 0% and maximum value theoretically 100%. Higher score means worse predicted outcome.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Population: Assessment of 10-year cardiovascular risk score based on the Framingham population derived algorithm.
  Minimum value 0% and maximum value theoretically 100%. Higher score means worse predicted outcome.
Measure: Mean (Standard Deviation); unit: % risk over 10 years
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
% risk over 10 years | -1.37 (5.68) | -1.23 (4.47)

11. Secondary Outcome: Change in QRisk Score
Description: Assessment of cardiovascular risk score based on the QRisk risk score. Minimum value 0% and maximum value theoretically 100%. Higher score means worse predicted outcome.
  Assessment of cardiovascular risk score based on the UK standardised using the QRISK2 algorithm (www.qrisk.org).
  Minimum value 0% and maximum value theoretically 100%. Higher score means worse predicted outcome.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Population: Assessment of cardiovascular risk score based on the UK standardised using the QRISK2 algorithm (www.qrisk.org).
  Minimum value 0% and maximum value theoretically 100%. Higher score means worse predicted outcome.
Measure: Mean (Standard Deviation); unit: % risk over 10-years
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
% risk over 10-years | -0.05 (2.64) | 0.2 (2.52)

12. Secondary Outcome: Change in Total Cholesterol to HDL Ratio
Description: Ratio of Total cholesterol to HDL from blood test for lipid profile. Change in the ratio of total cholesterol to HDL cholesterol ratio as assessed though cholesterol blood test. Negative value suggests an improvement.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Population: Change in the ratio of total cholesterol to HDL cholesterol ratio as assessed though cholesterol blood test. Negative value suggests an improvement.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
ratio | -0.11 (0.66) | -0.04 (0.55)

13. Secondary Outcome: Change in LDL Cholesterol
Description: Bloods for lipid profile. Change in the level of LDL cholesterol as assessed though cholesterol blood test. Negative value for change suggests an improvement.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Population: Change in the level of LDL cholesterol as assessed though cholesterol blood test. Negative value for change suggests an improvement.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
mmol/L | -0.2 (0.77) | -0.16 (0.68)

14. Secondary Outcome: Change in Glucose Levels
Description: Fasting glucose bloods. This is an assessment for presence of diabetes and control of blood sugar levels on the day of the test.
  Change in the blood glucose level as measure on the day of the visit as a measure of blood sugar level. Negative value would suggest an improvement.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Population: Change in the blood glucose level as measure on the day of the visit as a measure of blood sugar level. Negative value would suggest an improvement.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
mmol/L | -0.27 (0.87) | -0.29 (0.87)

15. Secondary Outcome: Change in hsCRP
Description: baseline and change in hsCRP blood test. hsCRP is measured through a blood test and is a marker of inflammation. Change in the hsCRP level though a blood test. Negative value suggests an improvement.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Population: Change in the hsCRP level though a blood test. Negative value suggests an improvement.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
mg/L | 0 (7.7) | -0.26 (8.19)

16. Secondary Outcome: Change in Physical Activity
Description: Lifestyle, quality of life and physical activity questionnaires. Questionnaires SF-36, EQ5D-3L, RPAQ
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Measure: Mean (Standard Deviation); unit: minutes per day over 5 days
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
minutes per day over 5 days | 8.45 (118.87) | 25.1 (132.85)

17. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure measured during sitting position
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
mmHg | -1.69 (13.91) | -3.18 (12.2)

18. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure measure during sitting position.
Time Frame: Assessed at Baseline visit, 3 months and 6 months; Month 6 reported
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
Number analyzed (Participants) | 183 | 194
mmHg | -2.08 (6.85) | -2.37 (6.41)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Care | Electronic Coaching Plus Standard Care
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/205
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/205
Other Adverse Events (participants affected / at risk) | 0/197 | 0/205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes